CLINICAL TRIAL: NCT05144009
Title: A Phase 2 Open-label Study of Loncastuximab Tesirine in Combination With Rituximab (Lonca-R) in Previously Untreated Unfit/Frail Patients With Diffuse Large B-cell Lymphoma (DLBCL) (LOTIS-9)
Brief Title: A Study of Loncastuximab Tesirine and Rituximab (Lonca-R) in Previously Untreated Unfit/Frail Participants With Diffuse Large B-cell Lymphoma (DLBCL)
Acronym: LOTIS-9
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The benefit-risk profile does not support continuation of the LOTIS-9 trial.
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-402-203; 2021-005312-57 (EudraCT Number); 2022-501601-12-00 (EU CTIS Number)
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Lymphoma; Loncastuximab Tesirine; Rituximab; Non-Hodgkin's lymphoma; Elderly; R-mini-CHOP; Geriatric Assessment; FIL Tool; Unfit; Frail
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, Non-Hodgkin | interventions — loncastuximab tesirine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A : Loncastuximab Tesirine + Rituximab (Lonca-R) (Experimental): Participants who are unfit (per sGA) will receive Lonca-R for 3 cycles. Participants who achieve a complete response (CR) will receive Lonca-R for 1 additional cycle. Participants who achieve a partial response (PR) will receive Lonca-R for 3 additional cycles.
  Lonca-R will be administered as rituximab 375 mg/m^2 on Day 1 of Cycle 1 and loncastuximab tesirine 150 µg/kg on Day 2 of Cycle 1. During Cycle 2, Lonca-R will be administered as rituximab* 375 mg/m^2 and loncastuximab tesirine 150 µg/kg on Day 1. For cycles 3 and beyond, Lonca-R will be administered as rituximab 375 mg/m^2 and loncastuximab tesirine 75 µg/kg on Day 1.
  *subcutaneous rituximab 1400mg/dose may be used during Cycle 2 and beyond
  Interventions: Drug: Loncastuximab Tesirine; Drug: Rituximab
- Cohort B : Loncastuximab Tesirine + Rituximab (Lonca-R) (Experimental): Participants who are frail (per sGA) or participants with cardiac comorbidities will receive Lonca-R for 3 cycles. Participants who achieve a CR will receive Lonca-R for 1 additional cycle. Participants who achieve a PR will receive Lonca-R for 3 additional cycles for a total of up to 6 cycles. Only participants enrolled in Cohort B, who achieve stable disease (SD) and deriving clinical benefit per the treating physician, may also receive Lonca-R for an additional 3 cycles.
  Lonca-R will be administered as rituximab 375 mg/m^2 on Day 1 of Cycle 1 and loncastuximab tesirine 150 µg/kg on Day 2 of Cycle 1. During Cycle 2, Lonca-R will be administered as rituximab* 375 mg/m^2 and loncastuximab tesirine 150 µg/kg on Day 1. For cycles 3 and beyond, Lonca-R will be administered as rituximab 375 mg/m^2 and loncastuximab tesirine 75 µg/kg on Day 1.
  *subcutaneous rituximab 1400mg/dose may be used during Cycle 2 and beyond
  Interventions: Drug: Loncastuximab Tesirine; Drug: Rituximab

INTERVENTIONS:
Drug: Loncastuximab Tesirine — Intravenous (IV) Infusion
  Other Names: Zynlonta; ADCT-402
Drug: Rituximab — Cycle 1 - Intravenous (IV) Infusion. Cycle 2+ - Intravenous (IV) Infusion or Subcutaneous (SC) Administration.

SUMMARY:
The main objective of the trial is to assess the efficacy and tolerability of Lonca-R in unfit and frail participants with previously untreated DLBCL.

DETAILED DESCRIPTION:
The primary objectives of this trial are shown below:

Cohort A: To assess the efficacy of a response-adapted treatment of Lonca-R in unfit participants with previously untreated DLBCL, high-grade B cell lymphoma (HGBCL), or Grade 3b follicular lymphoma (FL).

Cohort B: To assess the tolerability and efficacy of a response-adapted treatment of Lonca-R in frail participants with previously untreated DLBCL, or HGBCL, or Grade 3b FL who are ineligible for standard R-mini-CHOP.

The simplified geriatric assessment (sGA) developed by the Fondazione Italiana Linfomi (FIL) identifies three distinct categories (fit, unfit, and frail) based on age, activities of daily living (ADL), instrumental activities of daily living (IADL) and the Cumulative Illness Rating Scale for Geriatrics (CIRS-G). Participants will be assigned to Cohort A (unfit) or B (frail) using the sGA.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of DLBCL, as defined by the 2016 World Health Organization (WHO) classification (including participants with DLBCL transformed from indolent lymphoma), or HGBCL, or Grade 3b FL.
* Measurable disease as defined by the 2014 Lugano Classification.
* Stages I-IV.
* ECOG PS 0-2; ECOG PS 3 allowed if decline in status is deemed related to lymphoma & felt to be potentially reversible by the treating physician.
* Adequate organ function as defined by screening laboratory values within the following parameters:

  1. Absolute neutrophil count (ANC) ≥1.0 x 10^3/µL (off growth factors at least 72 hours).
  2. Platelet count ≥75 x 10^3/µL without transfusion in the past 7 days.
  3. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and gamma glutamyl transferase (GGT) ≤2.5 x the upper limit of normal (ULN).
  4. Total bilirubin ≤1.5 x ULN (participants with known Gilbert's syndrome may have a total bilirubin up to ≤3 x ULN).
  5. Calculated creatinine clearance >30 mL/min by the Cockcroft and Gault equation.

Note: A laboratory assessment may be repeated a maximum of two times during the screening period to confirm eligibility.

* Women of childbearing potential (WOCBP) must agree to use a highly effective method of contraception from the time of giving informed consent until at least 12 months after the last dose of study treatment. Men with female partners who are of childbearing potential must agree to use a condom when sexually active or practice total abstinence from the time of the first dose until at least 7 months after the participant receives his last dose of study treatment.

Inclusion Criteria specific for Cohort A:

* Unfit as defined by the simplified geriatric assessment (sGA). Includes all of the following:

  1. Aged ≥80 years
  2. ADL score of 6
  3. IADL score of 8
  4. CIRS-G: no score of 3-4 and <5 scores of 2

Inclusion Criteria specific for Cohort B:

* Frail as defined by sGA:

  1. Aged ≥80 years
  2. ADL score of <6 and/or
  3. IADL score of <8 and/or
  4. CIRS-G: ≥1 score of 3-4 and/or >5 scores of 2 OR
* Aged ≥65 - <80 with at least one of the following cardiac comorbidities that make anthracycline-containing regimens inadvisable as determined by the investigator.

  1. Left ventricular ejection fraction (LVEF) ≥30 to <50%
  2. History of myocardial infarction within 6 months prior to screening
  3. Ischemic heart disease
  4. History of stroke within 12 months prior to screening

Exclusion Criteria:

* Known history of hypersensitivity to or positive serum human anti-drug antibody to a cluster of differentiation 19 (CD19) antibody.
* Previous therapy for DLBCL, HGBCL, or Grade 3b FL (with exception of corticosteroid course for symptom management of less than 14 days).
* Previous therapy with loncastuximab tesirine and rituximab for any indication.
* Known history of hypersensitivity to any component of study treatment (loncastuximab tesirine and rituximab)
* Human immunodeficiency virus (HIV) seropositive with any of the following:

  1. CD4+ T-cell (CD4+) counts <350 cells/µL
  2. Acquired immunodeficiency syndrome (AIDS) - defining opportunistic infection within 12 months prior to screening
  3. Not on anti-retroviral therapy, or on anti-retroviral therapy for <4 weeks at the time of screening
  4. HIV viral load ≥400 copies/mL
* Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy or with detectable HBV viral load.
* Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load.
* History of Stevens-Johnson syndrome or toxic epidermal necrolysis.
* Lymphoma with active central nervous system involvement at the time of screening, including leptomeningeal disease.
* Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath).
* Major surgery, radiotherapy, chemotherapy, or other anti-neoplastic therapy within 14 days prior to start of study drug (Cycle 1 Day 1 [C1D1]), except shorter if approved by the Sponsor.
* Use of any other experimental medication within 14 days prior to start of study drug (C1D1).
* Received live vaccine within 4 weeks of C1D1.
* Congenital long QT syndrome or a corrected Fridericia correction of the QT measure (QTcF) interval of >480 ms at screening (unless secondary to pacemaker or bundle branch block).
* Active second primary malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's Medical monitor and Investigator agree, and document should not be exclusionary.
* Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgment, make the participant inappropriate for study participation or put the participant at risk.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (29):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Winthrop P. Rockefeller Cancer Institute, Little Rock, Arkansas
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - USOR - Illinois Cancer Specialists - Niles, Niles, Illinois
  - Leonard Lawson Cancer Center, Pikeville, Kentucky
  - Cancer Care Specialists - Nevada, Reno, Nevada
  - New York Cancer & Blood Specialists - New Hyde Park, Babylon, New York
  - New York Cancer & Blood Specialists - Babylon Medical Oncology, Port Jefferson, New York
  - Novant Health Cancer Specialists - Charlotte, Charlotte, North Carolina
  - USOR - Oncology Hematology Care - Kenwood, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio Health - Research and Innovation Institute, Columbus, Ohio
  - Willamette Valley Cancer Institute and Research Center - Eugene, Eugene, Oregon
  - Reading Hospital - Tower Health, Reading, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - USOR - Texas Oncology - Presbyterian Cancer Center Dallas, Dallas, Texas
  - USOR - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - USOR - Texas Oncology - San Antonio, San Antonio, Texas
  - Texas Oncology Northeast Texas - Tyler, Tyler, Texas
  - Blue Ridge Cancer Care - Blacksburg, Blacksburg, Virginia
  - USOR - Virginia Cancer Specialists - Gainesville Office, Gainesville, Virginia
  - Virginia Cancer Institute - West End, Richmond, Virginia
  - USOR - Virginia Oncology Associates, Virginia Beach, Virginia
  - Kadlec Clinic - Hematology and Oncology, Richland, Washington
  - USOR - Northwest Cancer Specialists, P.C. dba Compass Oncology - Vancouver Cancer Center, Vancouver, Washington
- Italy (3):
  - Ospedaliera Santi Antonio E Biagio E Cesare Arrigo-SC Ematologia, Alessandria
  - Azienda Socio Sanitaria Territoriale (ASST) degli Spedali Civili di Brescia, Brescia
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
- Hospital Español Auxilio Mutuo, San Juan, Puerto Rico
- Spain (8):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Arnau de Vilanova, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 41 participants were enrolled in the Unites States and Spain between June 2022 and January 2024.
Groups:
- Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R): Unfit participants (per simplified geriatric assessment [sGA]) received Lonca-R for 3 cycles (each treatment cycle was 3 weeks). A response-adapted approach was implemented, where participants achieving complete response (CR) after 3 cycles received 1 additional cycle (4 cycles total), and those with partial response (PR) after 3 cycles received additional cycles based on their cohort assignment (6 cycles total).
  Loncastuximab tesirine was administered as an intravenous (IV) infusion on Day 2 of Cycle 1 and Day 1 (prior to rituximab administration) of subsequent cycles. Participants received 150 μg/kg loncastuximab tesirine for 2 cycles, followed by 75 μg/kg loncastuximab tesirine for subsequent cycles. Rituximab was administered as an IV infusion on Day 1 of each cycle at a dose of 375 mg/m^2.
- Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R): Frail participants (per sGA) or participants with cardiac comorbidities received Lonca-R for 3 cycles (each treatment cycle was 3 weeks). A response-adapted approach was implemented, where participants achieving CR after 3 cycles received 1 additional cycle (4 cycles total), and those with PR or stable disease (SD) (Cohort B only) after 3 cycles received additional cycles based on their cohort assignment (6 cycles total).
  Loncastuximab tesirine was administered as an IV infusion on Day 2 of Cycle 1 and Day 1 (prior to rituximab administration) of subsequent cycles. Participants received 150 μg/kg loncastuximab tesirine for 2 cycles, followed by 75 μg/kg loncastuximab tesirine for subsequent cycles. Rituximab was administered as an IV infusion on Day 1 of each cycle at a dose of 375 mg/m^2.
Period: Overall Study
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Started | 17 | 24
Completed | 0 | 0
Not Completed | 17 | 24
Not completed — Lost to Follow-up | 0 | 1
Not completed — Study Termination by the Sponsor | 11 | 11
Not completed — Disease Progression | 1 | 0
Not completed — Participant Decision | 0 | 2
Not completed — Death | 5 | 10

BASELINE CHARACTERISTICS:
Population: All-Treated Population: all participants who received at least 1 dose of study drug.
Groups:
- Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R): Unfit participants (per sGA) received Lonca-R for 3 cycles (each treatment cycle was 3 weeks). A response-adapted approach was implemented, where participants achieving CR after 3 cycles received 1 additional cycle (4 cycles total), and those with PR after 3 cycles received additional cycles based on their cohort assignment (6 cycles total).
  Loncastuximab tesirine was administered as an IV infusion on Day 2 of Cycle 1 and Day 1 (prior to rituximab administration) of subsequent cycles. Participants received 150 μg/kg loncastuximab tesirine for 2 cycles, followed by 75 μg/kg loncastuximab tesirine for subsequent cycles. Rituximab was administered as an IV infusion on Day 1 of each cycle at a dose of 375 mg/m^2.
- Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R): Frail participants (per sGA) or participants with cardiac comorbidities received Lonca-R for 3 cycles (each treatment cycle was 3 weeks). A response-adapted approach was implemented, where participants achieving CR after 3 cycles received 1 additional cycle (4 cycles total), and those with PR or SD (Cohort B only) after 3 cycles received additional cycles based on their cohort assignment (6 cycles total).
  Loncastuximab tesirine was administered as an IV infusion on Day 2 of Cycle 1 and Day 1 (prior to rituximab administration) of subsequent cycles. Participants received 150 μg/kg loncastuximab tesirine for 2 cycles, followed by 75 μg/kg loncastuximab tesirine for subsequent cycles. Rituximab was administered as an IV infusion on Day 1 of each cycle at a dose of 375 mg/m^2.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R) | Total
Number analyzed (Participants) | 17 | 24 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.1 (3.48) | 80.0 (7.07) | 81.7 (6.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 14 | 20 | 34
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 16 | 22 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: CR Rate
Description: Defined as percentage of participants with a best overall response (BOR) of CR as determined by the Investigator according to the 2014 Lugano Classification criteria.
  CR was defined as achieving:
  * Complete metabolic response for positron emission tomography (PET)-computed tomography (CT) OR
  * Complete radiologic response (target node regress to <1.5 cm, no non-measured lesions, no organ enlargement, no new lesions and normal bone marrow morphology) for CT if disease was not fluorodeoxyglucose (FDG)-avid at baseline.
Time Frame: Up to a maximum of 17.1 months
Population: All-Treated Population: All participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 17 | 24
percentage of participants | 52.9 [27.8 to 77.0] | 41.7 [22.1 to 63.4]

2. Primary Outcome: Cohort B: Percentage of Participants Who Completed 4 Cycles of Treatment
Description: Defined by the number of participants who completed a total of 4 cycles of therapy divided by the total number of participants * 100.
Time Frame: Up to 12 weeks (3 week cycle length)
Population: All-Treated Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 24
percentage of participants | 33.3

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Defined as the percentage of participants who achieved either CR or PR as BOR as determined by Investigator according to the 2014 Lugano Classification criteria.
  CR was defined as achieving:
  * Complete metabolic response for PET-CT OR
  * Complete radiologic response (target node regress to <1.5 cm, no non-measured lesions, no organ enlargement, no new lesions and normal bone marrow morphology) for CT if disease was not FDG-avid at baseline.
  PR was defined as achieving:
  * Partial metabolic response (findings indicate residual disease) for PET-CT OR
  * Partial remission (>50% decrease in target measurable nodes, regression/ absence/ no increase of non-measured lesions, spleen regressed by >50% in length and no new lesions) for CT if disease was not FDG-avid at baseline.
Time Frame: Up to a maximum of 17.1 months
Population: All-Treated Population: All participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 17 | 24
percentage of participants | 94.1 [71.3 to 99.9] | 66.7 [44.7 to 84.4]

4. Secondary Outcome: 2-year Progression-free Survival (PFS)
Description: PFS was defined as the time from first dose of study drug until the first date of either disease progression (PD) or death due to any cause. The 2-year PFS was defined as the percentage of participants that were PFS event-free at 2 years per investigator assessment with 95% confidence interval (CI) estimated using Kaplan-Meier method.
Time Frame: 2 years
Population: All-Treated Population: All participants who received at least 1 dose of study drug. No data was collected for this endpoint due to study early termination.
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: 3-year Overall Survival (OS)
Description: OS was defined as the time from randomization date until death due to any cause. The 3-year OS was defined as the percentage of participants that were OS event-free at 3 years with 95% CI estimated using Kaplan-Meier method.
Time Frame: 3 years
Population: as for outcome 4
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Response (DoR)
Description: Defined for participants with CR or PR only as the interval between the date of initial documentation of a response and the date of the first documented progressive disease (based on radiographic or clinical progression at end of study or death due to any cause, whichever occurred first) per investigator assessment with 95% CI estimated using Kaplan-Meier method.
  CR was defined as achieving:
  * Complete metabolic response for PET-CT OR
  * Complete radiologic response (target node regress to <1.5 cm, no non-measured lesions, no organ enlargement, no new lesions and normal bone marrow morphology) for CT if disease was not FDG-avid at baseline.
  PR was defined as achieving:
  * Partial metabolic response (findings indicate residual disease) for PET-CT OR
  * Partial remission (>50% decrease in target measurable nodes, regression/ absence/ no increase of non-measured lesions, spleen regressed by >50% in length and no new lesions) for CT if disease was not FDG-avid at baseline.
Time Frame: Up to a maximum of 17.1 months
Population: All-Treated Population: All participants who received at least 1 dose of study drug. Inclusive of participants who were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 17 | 24
months | 5.49 [2.27 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | NA [NA to NA] — Median and confidence intervals were not calculable due to insufficient event data occurring near the median.

7. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product. A TEAE was defined as an AE that occurred or worsened in the period extending from the first dose of study drug to 15 weeks after the last dose of study drugs in this study or start of a new anticancer therapy, whichever was earlier. A serious AE (SAE) was defined as an AE that resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or an important medical event. A severe AE was defined as Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade 3 (severe) or above.
  Clinically significant changes in safety laboratory variables, vital signs, physical examinations, and Eastern Cooperative Oncology Group performance score were recorded as AEs.
Time Frame: Up to approximately 8 months
Population: All-Treated Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 17 | 24
Participants
  Any TEAEs | 17 | 23
  Any CTCAE Grade 3 or Higher TEAEs | 13 | 18
  Any Serious TEAEs | 13 | 16

8. Secondary Outcome: Maximum Observed Concentration (Cmax) of Conjugated Antibody
Description: Pharmacokinetic (PK) was assessed by a central laboratory using validated bioanalytical methods. Analysis considered model development for conjugated antibodies and total antibodies only, as pre-specified in protocol section 9.9.
Time Frame: Cycle 1 Day 2: predose (preferably within 2 h prior to start of infusion) and at the end (within -5 to +10 min) of loncastuximab tesirine infusion; Cycles 2-6 Day 1 predose and at the end of loncastuximab tesirine infusion (3 week cycle length)
Population: PK Population: All participants who received study drug and have at least 1 pre-(Cycle 1 Day 1) and 1 post-dose valid PK assessment. Inclusive of only participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 17 | 18
ng/mL
  Cycle 1 | 1667 (274) | 1788 (52.2)
  Cycle 2: number analyzed (Participants) | 16 | 18
  Cycle 2 | 2461 (65.2) | 2353 (30.5)
  Cycle 3: number analyzed (Participants) | 15 | 14
  Cycle 3 | 1456 (40.6) | 1407 (29.6)
  Cycle 4: number analyzed (Participants) | 15 | 7
  Cycle 4 | 1581 (28.6) | 1163 (59.4)
  Cycle 5: number analyzed (Participants) | 7 | 3
  Cycle 5 | 1377 (18.2) | 1700 (15.2)
  Cycle 6: number analyzed (Participants) | 3 | 3
  Cycle 6 | 1087 (28.2) | 617 (83.9)

9. Secondary Outcome: Cmax of Total Antibody
Description: PK was assessed by a central laboratory using validated bioanalytical methods. Analysis considered model development for conjugated antibodies and total antibodies only, as pre-specified in protocol section 9.9.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 17 | 21
ng/mL
  Cycle 1 | 2751 (59.4) | 1971 (115)
  Cycle 2: number analyzed (Participants) | 16 | 19
  Cycle 2 | 3270 (68.6) | 2746 (33.5)
  Cycle 3: number analyzed (Participants) | 15 | 14
  Cycle 3 | 2010 (49.0) | 1834 (32.6)
  Cycle 4: number analyzed (Participants) | 15 | 7
  Cycle 4 | 2044 (44.8) | 1362 (56.8)
  Cycle 5: number analyzed (Participants) | 7 | 3
  Cycle 5 | 1874 (36.0) | 1799 (25.9)
  Cycle 6: number analyzed (Participants) | 3 | 3
  Cycle 6 | 1466 (19.1) | 1175 (110)

10. Secondary Outcome: Trough Concentration (Ctrough) of Conjugated Antibody
Description: as for outcome 9
Time Frame: Cycle 1 Day 2: predose (preferably within 2 h prior to start of infusion); Cycles 2-6 Day 1 predose (3 week cycle length)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 15 | 17
ng/mL
  Cycle 1 | 324 (30.7) | 215 (142)
  Cycle 2: number analyzed (Participants) | 15 | 14
  Cycle 2 | 548 (35.6) | 449 (70.3)
  Cycle 3: number analyzed (Participants) | 15 | 7
  Cycle 3 | 411 (53.8) | 479 (35.1)
  Cycle 4: number analyzed (Participants) | 7 | 3
  Cycle 4 | 391 (25.4) | 436 (32.1)
  Cycle 5: number analyzed (Participants) | 3 | 3
  Cycle 5 | 353 (24.0) | 453 (34.8)
  Cycle 6: number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Ctrough of Total Antibody
Description: as for outcome 9
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 15 | 18
ng/mL
  Cycle 1 | 503 (75.1) | 413 (56.9)
  Cycle 2: number analyzed (Participants) | 15 | 14
  Cycle 2 | 805 (68.5) | 650 (70.2)
  Cycle 3: number analyzed (Participants) | 15 | 7
  Cycle 3 | 619 (75.9) | 645 (31.5)
  Cycle 4: number analyzed (Participants) | 7 | 3
  Cycle 4 | 633 (69.1) | 627 (26.9)
  Cycle 5: number analyzed (Participants) | 3 | 3
  Cycle 5 | 509 (31.8) | 658 (40.2)
  Cycle 6: number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Confirmed Positive Anti-Drug Antibody (ADA) Response
Description: Detection of ADAs against loncastuximab tesirine was performed by using a screening assay for identification of antibody positive samples/participants and a confirmation assay. A participant was considered to have an ADA response if ADA sample was positive at any pre-specified, post-treatment timepoint.
Time Frame: Cycle 1 Day 2 pre-dose (preferably within 2 h prior to start of infusion) then Day 1 pre-dose of Cycles 2, 4, and 6 (3 week cycle length)
Population: Immunogenicity Population: All participants who received study drug and had at least 1 valid anti-drug antibody assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 17 | 24
Participants | 0 | 0

13. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) Subscale and Composite Scores
Description: The following score ranges were possible for the FACT-Lym subscale and composite scores, with higher scores indicating better quality of life/outcome: 0 to 28 for physical well-being, social/family well-being, and functional well-being; 0 to 24 for emotional well-being; 0 to 60 for lymphoma subscale score; 0 to 116 for FACT-Lym trial outcome index; 0 to 108 for FACT-G total score; and 0 to 168 for FACT-Lym Total. An increase in subscale/composite scores from Baseline indicated better quality of life/outcome.
Time Frame: Baseline and End of Treatment Visit (a maximum of 19 weeks)
Population: Patient-reported Outcomes Population: All participants who received at least one dose of study treatment and completed at least one questionnaire at Baseline and at one post Baseline visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
Number analyzed (Participants) | 10 | 12
score on a scale
  Physical Well-being Subscale | -5.70 (4.811) | -1.55 (4.793)
  Social/family Well-being Subscale | 0.52 (1.895) | 1.22 (5.675)
  Emotional Well-being Subscale | 2.10 (4.280) | -0.95 (2.396)
  Functional Well-being Subscale | -3.63 (3.860) | -1.44 (6.675)
  Lymphoma Subscale: number analyzed (Participants) | 9 | 12
  Lymphoma Subscale | -4.29 (10.577) | -0.08 (8.385)
  FACT-Lymphoma Trial Outcome Index: number analyzed (Participants) | 9 | 12
  FACT-Lymphoma Trial Outcome Index | -11.99 (16.188) | -3.08 (12.452)
  FACT-G | -6.71 (11.889) | -2.72 (10.649)
  FACT-Lymphoma: number analyzed (Participants) | 9 | 12
  FACT-Lymphoma | -8.71 (18.267) | -2.81 (14.953)

ADVERSE EVENTS:
Time Frame: All cause mortality: up to a maximum of 17.1 months; serious and other adverse events: up to approximately 8 months
Description: All-Treated Population: All participants who received at least 1 dose of study drug.
Arm/Group | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R)
All-Cause Mortality (participants affected / at risk) | 5/17 | 10/24
Serious Adverse Events (participants affected / at risk) | 13/17 | 16/24
Other Adverse Events (participants affected / at risk) | 17/17 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) (N=17) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R) (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 5 (5)
Sepsis (Infections and infestations) | 2 (3) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Loncastuximab Tesirine + Rituximab (Lonca-R) (N=17) | Cohort B: Loncastuximab Tesirine + Rituximab (Lonca-R) (N=24)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pericardial effusion (Cardiac disorders) | 5 (6) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (9) | 10 (10)
Oedema peripheral (General disorders) | 8 (11) | 7 (7)
Face oedema (General disorders) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Generalised oedema (General disorders) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 2 (3) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (3) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3)
Cytomegalovirus gastritis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 3 (4) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 3 (3)
Weight increased (Investigations) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (6) | 3 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (5) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin weeping (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, the objectives of the study could not be fully assessed (e.g. overall survival). The median duration of follow-up for all participants was limited because of early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT05144009/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT05144009/SAP_001.pdf